CLINICAL TRIAL: NCT03626363
Title: Randomized, Active-Control Study to Determine the Effect of Mindfulness-Based Stress Reduction on Sympathetic Activity and Arterial Stiffness
Brief Title: Mindfulness and Neural Cardiovascular Control in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan Technological University (Other)
Collaborators: Emory University (Other); Texas Tech University (Other); Purdue University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M1690; 1R15HL140596-01 (NIH)
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Elevated Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): An 8-week program specifically designed to improve mindfulness and to reduce stress.
  Interventions: Behavioral: Stress Management
- Stress Management Education (Active Comparator): An 8-week program specifically designed to provide education about stress responses in humans, and as an active control for Mindfulness-Based Stress Reduction studies.
  Interventions: Behavioral: Stress Management

INTERVENTIONS:
Behavioral: Stress Management — An eight week stress reduction course.

SUMMARY:
This study evaluates the impact of mindfulness-based stress reduction (MBSR) on sympathetic nerve activity and arterial stiffness. The investigator's central hypothesis is that MBSR will reduce sympathetic activity and arterial stiffness.

DETAILED DESCRIPTION:
This study will recruit male and female subjects with elevated blood pressure who will participate in a randomized, active control study to examine the impact of mindfulness-based stress reduction (MBSR) on blood pressure, muscle sympathetic nerve activity and arterial stiffness. The study will utilize established techniques for assessing blood pressure patterns (24-hour ambulatory monitoring), peripheral sympathetic activity (microneurography) and vascular stiffness (applanation tonometry) in humans. This study includes a stress management education class for the active control.

ELIGIBILITY:
Inclusion Criteria:

* Seated systolic blood pressure >119 mmHg and/or diastolic blood pressure >79 mmHg
* Body mass index <30 kg/m2

Exclusion Criteria:

* Smokers
* Diabetes
* Pregnant women
* History of autonomic dysfunction
* Cardiovascular medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Durocher, PhD, Principal Investigator — Purdue University Northwest Biological Sciences
Locations (1):
- Purdue University Northwest, Hammond, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We screened 180 potential participants for this study between the fall of 2018 through the fall of 2022.
Groups:
- Mindfulness-Based Stress Reduction: An eight week course designed to increase mindfulness and to decrease stress. Participants met with an MBSR expert once each week for 2.5 hours and had at-home practice assignments for 45 minutes per day which included mindfulness, breathing, and gently yoga exercises.
- Stress Management Education: An eight week stress education course designed to be an active control for mindfulness-based stress reduction studies. Participants met for 2.5 hours each week to be educated about stress responses, benefits of gentle resistance training, and other topics such as the benefits of volunteering. Participants completed at-home sessions for 45-minutes each day that included reading from "Why Zebra's Don't Get Ulcers" and they could also perform gentle resistance training with a resistance band kit that was provided.
Period: Overall Study
Arm/Group | Mindfulness-Based Stress Reduction | Stress Management Education
Started | 27 | 25
Completed | 18 | 18
Not Completed | 9 | 7
Not completed — Protocol Violation | 4 | 0
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Mindfulness-Based Stress Reduction: An eight week course specifically designed to improve mindfulness and to reduce stress.
- Stress Management Education: An eight week program specifically designed to provide education about stress responses in humans, and as an active control for Mindfulness-Based Stress Reduction studies.
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Stress Reduction | Stress Management Education | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 26 | 25 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (7) | 23 (3) | 25 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 21 | 21 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 10 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52
muscle sympathetic nerve activity (MSNA) [Mean (Standard Deviation); unit: bursts per minute] — Population: Obtaining clear recordings of muscle sympathetic nerve activity is difficult and we cannot always obtain a clear signal with distinct bursts in all participants. Some participants elect not to have this measurement performed because it is invasive and can cause some temporary discomfort.
  bursts per minute
    number analyzed (Participants) | 18 | 14 | 32
    (all) | 19.6 (8.8) | 17.7 (5.9) | 18.8 (7.6)
Carotid-femoral pulse wave velocity (arterial stiffness) [Mean (Standard Deviation); unit: meters per second] | 5.55 (0.81) | 5.38 (0.82) | 5.47 (0.81)
Nocturnal systolic blood pressure dipping (%) [Mean (Standard Deviation); unit: Percent dipping vs. wakefulness average] — Population: We have only included participants with more than 80% successful wake and sleep measurements of ambulatory blood pressure. Three readings an hour were taken during wakefulness and two readings per hour were taken during sleep. Some participants did not keep the ambulatory monitor on during the entire recording period and others did not have the required percentage of successful recordings.
  Percent dipping vs. wakefulness average
    number analyzed (Participants) | 20 | 15 | 35
    (all) | 12.65 (7.13) | 12.66 (4.69) | 12.66 (6.12)

OUTCOME MEASURES:

1. Primary Outcome: Muscle Sympathetic Nerve Activity
Description: Direct recordings of muscle sympathetic nerve activity from the peroneal nerve using microneurography. Sympathetic bursts that were at least three times higher than baseline noise were evaluated by a trained investigator and quantified as bursts per minute. The investigator was blinded to the condition and whether the data was pre or post until after all data was collected and analyzed.
Time Frame: Data reported is the change in the mean value from before to after the 8 week intervention (i.e. pre to post).
Population: We had 21 participants in the spring of 2020 with excellent success on baseline nerve recordings, but with COVID-19 restrictions we were not allowed to bring any participants into the laboratory for post testing. This resulted in the limited sample size of 5 participants in each arm with excellent muscle sympathetic nerve recordings both before and after the 8-week interventions.
Measure: Mean (Standard Error); unit: bursts per minute
Arm/Group | Mindfulness-Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 5 | 5
bursts per minute | -2 (2) | -1 (2)
Statistical Analysis 1: Comparison: Mindfulness-Based Stress Reduction vs Stress Management Education; Repeated measures analysis of variance with 2 groups (MBSR and SME) and 2 time points (Pre vs. Post). Outcome data reported is the change in the mean number of bursts per minute of muscle sympathetic nerve activity (MSNA) from pre to post; Test type: Superiority — We sought to have up to 20 participants complete each group so that we could have a statistical power of 0.89 to detect about a 4 burst per minute difference with an alpha of 0.05. We would have had sympathetic nerve data on up to 18 more of the 21 participants that we were not allowed to post-test in the spring of 2020 due to COVID-19 restrictions; p = 0.51, ANOVA; Mean Difference (Net) = -2

2. Secondary Outcome: Arterial Stiffness
Description: Carotid-femoral pulse wave velocity using applanation tonometry. A SphygmoCor system was used to gait pulse waves from a tonometer to the R-wave of a 3-lead ECG and carotid to femoral pulse wave velocity was evaluated in meters per second. A higher value indicates more arterial stiffness in the aorta, and a lower value indicates less stiffness in the aorta.
Time Frame: Data reported is the change in the mean value from before to after the 8 week intervention (i.e. pre to post).
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- Mindfulness-Based Stress Reduction: An eight week program specifically designed to improve mindfulness and to reduce stress.
Arm/Group | Mindfulness-Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 10 | 12
meters per second | -0.04 (0.94) | -0.31 (0.72)
Statistical Analysis 1: Comparison: Mindfulness-Based Stress Reduction vs Stress Management Education; Repeated measures analysis of variance with 2 groups (MBSR and SME) and 2 time points (Pre vs. Post). Outcome data reported is the change in carotid-to-femoral pulse wave velocity in meters per second from pre to post. We had 21 participants in the spring of 2020 that were were not allowed to bring into the laboratory for post testing during COVID-19 restrictions which led to our limited sample size; Test type: Superiority — To detect a 0.5 meter per second change in carotid-to-femoral pulse wave velocity with at least 80% power with an alpha of 0.05 we should have had at least 12 participants complete measurements in each group (MBSR and SME). We fell a little short of that in the MBSR group and met the 12 participants in the SME group. The number of participants we were able to study from pre to post was limited by COVID-19 restrictions; p = 0.25, ANOVA; Mean Difference (Net) = -0.2

3. Other Pre Specified Outcome: Nocturnal Blood Pressure Dip
Description: Change in systolic nocturnal blood pressure during sleep when compared to wakefulness. We used ambulatory blood pressure monitors set to record blood pressures every 30 minutes while the participant was sleeping and every 20 minutes while they were awake for a 24-hour period once before and once after the 8-week intervention. Values reported are the percentage of systolic arterial pressure dipping during sleep compared to wakefulness before vs. after the 8 week intervention.
Time Frame: Data reported is the change in the mean value from before to after the 8 week intervention (i.e. pre to post).
Population: Repeated measures analysis of variance with 2 groups (MBSR and SME) and 2 time points (pre vs. post). Outcome data reported is the change in the mean nighttime systolic blood pressure dipping from pre to post as a percentage. We had 21 participants in the spring of 2020 that we were not allowed to bring into the laboratory for post-testing due to COVID-19 restrictions. We were only able to have participants in that largest cohort complete questionnaire data.
Measure: Mean (Standard Error); unit: percent dipping
Arm/Group | Mindfulness-Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 3 | 4
percent dipping | -3 (5) | 1 (6)

ADVERSE EVENTS:
Time Frame: Participants were randomized into an 8-week mindfulness-based stress reduction OR 8-week stress management education intervention. We pre-tested participants within a week of starting the interventions, and then post-tested them within a week of completing the interventions. Thus, each participant was monitored for a period of 10 weeks.
Arm/Group | Mindfulness-Based Stress Reduction | Stress Management Education
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/25

LIMITATIONS AND CAVEATS:
In spring 2020 we had 21 participants enrolled, and we shifted the MBSR and SME courses to Zoom for the final 4 weeks of each intervention. We were able to send out questionnaires to participants for post testing, but we were not allowed to post-test anyone in the lab for our three specific aims related to blood pressure dipping, MSNA, or arterial stiffness due to COVID-19 restrictions. The original PI moved to a new position in the summer of 2020 which provided some additional complications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT03626363/Prot_SAP_000.pdf
  • Informed Consent Form: Purdue Consent Form (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT03626363/ICF_001.pdf
  • Informed Consent Form: Michigan Tech Original Consent Form (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT03626363/ICF_002.pdf